CLINICAL TRIAL: NCT06696729
Title: External Application of Traditional Chinese Medicine Mirabilite for the Prevention of Incisional Complications and Promotion of Gastrointestinal Function Recovery in Gastrointestinal Surgery
Brief Title: External Application of Mirabilite to Promote Recovery in Patients After Gastrointestinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanchang University (Other)
Responsible Party: Principal Investigator, Taiyuan Li, professor, Nanchang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIT2024323
Record Dates: First submitted 2024-11-13; First posted 2024-11-20 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Gastrointestinal Surgery; Mirabilite; Surgical Site Infection; Postoperative Gastrointestinal Dysfunction
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mirabilite Application Group (Experimental): Participants will receive a 500-gram external application of Mirabilite on the abdominal incision site, replaced regularly to maintain efficacy.
  Interventions: Procedure: Topical Mirabilite Application for Postoperative Gastrointestinal Patients
- Standard Care Group (Sham Comparator): Participants will receive standard postoperative care with regular sterile dressing changes, without additional topical treatments.
  Interventions: Procedure: Standard Postoperative Care for Gastrointestinal Patients

INTERVENTIONS:
Procedure: Topical Mirabilite Application for Postoperative Gastrointestinal Patients — Participants in this group will receive an external application of 500 grams of Mirabilite (sodium sulfate decahydrate) beginning on postoperative day 1. The Mirabilite will be wrapped in a double layer of gauze and placed on top of the sterile dressing over the patient's abdominal incision, with the gauze bag secured by an abdominal binder. The application will be regularly replaced when it becomes damp and hardened to maintain continuous efficacy.
  Arms: Mirabilite Application Group
Procedure: Standard Postoperative Care for Gastrointestinal Patients — Participants in this group will receive standard postoperative care without the application of Mirabilite or any alternative topical treatment. Their surgical sites will be kept dry and clean, with regular sterile dressing changes as part of standard care protocols.
  Arms: Standard Care Group

SUMMARY:
This study evaluates the efficacy and safety of topical Mirabilite (sodium sulfate) application for managing postoperative outcomes in patients undergoing gastrointestinal cancer surgery. Conducted at the First Affiliated Hospital of Nanchang University, this randomized controlled trial assesses Mirabilite's potential to mitigate postoperative complications, including surgical site infections and abdominal distention, and to expedite the recovery of gastrointestinal function. Participants are randomly assigned to either a Mirabilite treatment group or a standard care control group. Follow-up assessments, extending up to five years, will examine incision healing, complication incidence, and metrics of gastrointestinal recovery to provide robust evidence on the clinical benefits of Mirabilite in surgical settings.

DETAILED DESCRIPTION:
This single-center randomized controlled trial investigates the efficacy of Mirabilite in enhancing postoperative outcomes for patients undergoing gastrointestinal surgery, with a specific focus on individuals receiving abdominal incisions for gastrointestinal malignancies. Abdominal surgeries often lead to complications such as incision fat liquefaction, surgical site infections (SSI), and postoperative gastrointestinal dysfunction, issues for which traditional treatment methods have shown limited success. This study aims to assess Mirabilite's potential therapeutic advantages in this context.

Mirabilite, a mineral widely used in traditional Chinese medicine, possesses properties that facilitate swelling reduction, pain relief, and tissue repair, attributed to its high osmotic pressure. Approximately 300 participants are randomly allocated to either a Mirabilite intervention group or a standard postoperative care group. In the intervention group, Mirabilite is applied topically to surgical incisions, with subsequent evaluations focusing on incision healing, gastrointestinal function recovery, and markers of inflammation.

Primary endpoints include incision healing duration, time to first flatus, SSI incidence, postoperative pain scores, and hospital length of stay. This trial seeks to substantiate the role of Mirabilite as a cost-effective and safe adjunct therapy for postoperative recovery in gastrointestinal surgery, with the potential to reduce hospital stays and mitigate complication rates.

ELIGIBILITY:
Inclusion Criteria:

* Underwent gastrointestinal surgery. Aged between 18 and 80 years. Provided signed informed consent.

Exclusion Criteria:

* Required unplanned surgical intervention within 30 days postoperatively. Presented with emergency conditions, such as bowel obstruction or gastrointestinal bleeding, or diagnosed with severe psychiatric disorders.

Underwent surgical procedures for advanced malignancies, including palliative or bypass surgeries.

Classified as American Society of Anesthesiologists (ASA) Physical Status > 3. Requested withdrawal from the study after enrollment. Demonstrated non-compliance or utilized mirabilite for fewer than three consecutive days.

Experienced unexpected discharge during the study period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Complications (%) | Within 30 days post-surgery
  The overall incidence of postoperative complications, including any adverse events directly related to the surgery.
Incidence of Surgical Site Infection (SSI) (%) | Within 30 days post-surgery
  The incidence rate of surgical site infections, categorized as superficial or deep infections at the incision site.
Time to First Flatus (Days) | 1 day after operation
  The duration in days from surgery to the first passage of flatus, indicating the resumption of gastrointestinal motility.

SECONDARY OUTCOMES:
C-Reactive Protein (CRP) Levels (mg/L) | Measured on postoperative days 1, 4, and 7.
  CRP levels as an inflammatory marker.
Visual Analog Scale (VAS) Pain Scores | Recorded on postoperative days 1, 2, and 3.
  Patient-reported pain levels on a 10-cm VAS scale (0 = no pain, 10 = worst pain).
Daily Drainage Volume (mL) | Measured daily from postoperative days 1 through 7.
  Total daily output from drainage tubes, indicating postoperative exudation and inflammation.
Postoperative Serum Protein Levels (g/L) | Measured on postoperative days 1 and 4.
  Serum protein levels, reflecting nutritional status and recovery.
Length of Postoperative Hospital Stay (Days) | 1 day after operation
  Total duration of hospital stay post-surgery.
Operative Time (Minutes) | Recorded on the day of surgery.
  Duration of the surgical procedure.
Incision Length (cm) | Measured on the day of surgery.
  Length of the surgical incision made during the procedure.
Surgical Type | Recorded on the day of surgery.
  Classification of the surgical procedure type
Intraoperative Blood Loss (mL) | Measured on the day of surgery.
  Total volume of blood lost during the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Ye ShanPing Dr. Ye, Study Chair — Department of General Surgery, The First Affiliated Hospital, Jiangxi Medical College, Nanchang University, Nanchang 330006, Jiangxi Province, China
Locations (1):
- the First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No